CLINICAL TRIAL: NCT01261091
Title: Stroke-Related Early Tracheostomy vs. Prolonged Orotracheal Intubation in Neurocritical Care Trial
Brief Title: Early Tracheostomy in Ventilated Stroke Patients
Acronym: SETPOINT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Julian Boesel, PD Dr.med., Attending Neurology, Director NCCU, Heidelberg University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: S-060/2009
Record Dates: First submitted 2010-12-15; First posted 2010-12-16 (Estimated); Last update posted 2014-04-24 (Estimated); Status verified 2014-04

CONDITIONS: Ischemic Stroke; Intracerebral Hemorrhage; Subarachnoid Hemorrhage
Keywords: Neurocritical Care; Ischemic Stroke; Intracerebral Hemorrhage; Subarachnoid Hemorrhage; Tracheostomy; Tracheotomy; Percutaneous Dilatative Tracheostomy; Weaning; Ventilation
MeSH Terms: conditions — Ischemic Stroke; Cerebral Hemorrhage; Subarachnoid Hemorrhage; Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Early Tracheostomy (Experimental): Patients randomized to early tracheostomy receive (preferably dilatative) tracheostomy within 3 days from intubation.
  Interventions: Procedure: Early Tracheostomy
- Prolonged Intubation (Active Comparator): Patients randomized to this arm will be tried to wean off the ventilator and get (an) extubation trial(s) if regarded feasible. In case of failure or non-feasibility, they receive tracheostomy between days 7 to 14 from intubation.
  Interventions: Procedure: Late Tracheostomy

INTERVENTIONS:
Procedure: Early Tracheostomy — Tracheostomy is performed as percutaneous dilatative tracheostomy by neurointensivists whenever possible. If anatomically or otherwise indicated, surgical tracheostomy is applied.
  Arms: Early Tracheostomy
Procedure: Late Tracheostomy — Tracheostomy is performed as percutaneous dilatative tracheostomy by neurointensivists whenever possible. If anatomically or otherwise indicated, surgical tracheostomy is applied.
  Arms: Prolonged Intubation

SUMMARY:
Patients with severe ischemic and hemorrhagic strokes, who require mechanical ventilation, have a particularly bad prognosis. If they require long-term ventilation, their orotracheal tube needs to be, like in any other intensive care patient, replaced by a shorter tracheal tube below the larynx. This so called tracheostomy might be associated with advantages such as less demand of narcotics and pain killers, less lesions in mouth and larynx, better mouth hygiene, safer airway, more patient comfort and earlier mobilisation. The best timepoint for tracheostomy in stroke, however, is not known. This study investigates the potential benefits of early tracheostomy in ventilated critically ill patients with ischemic or hemorrhagic stroke.

DETAILED DESCRIPTION:
Background: Tracheostomy is a common procedure in critical care patients. Advantages of a short tracheal tube compared to a long orotracheal one are the avoidance of laryngeal lesions and sinusitis, facilitation of nursing care and physiotherapy and the reduction of analgosedatives. The optimal point in time for tracheostomy is still unknown, but it is commonly done not later than 2-3 weeks and after one or several failed extubation trials. Studies in different sets of critical care patients have suggested additional advantages of early tracheostomy: less pneumonias and other complications, more patient comfort, less analgosedation, shorter duration of ventilation and of ICU stay. These questions have not been looked at in non-traumatic neurocritical care patients, although these might have a special weaning benefit by early tracheostomy, being mainly compromised in securing their airway, but not in breathing.

Method: Non-traumatic Neurocritical care patients with ischemic strokes, intracerebral hemorrhage or subarachnoid hemorrhage so severly affected that 2 weeks of ventilation need are estimated, are principally eligible for the study. After randomization, one group receives tracheostomy within the first 3 days after intubation. The other group stays orotracheally intubated and is either weaned and extubated or receives tracheostomy within 7 to 14 days after intubation. Tracheostomy is done as percutaneous dilatation by neurologists.

ELIGIBILITY:
Inclusion Criteria:

* age > 18 years
* informed consent from legal representative
* non-traumatic cerebrovascular disease
* Estimated ventilation need for at least 2 weeks

Exclusion Criteria:

* age < 18 years
* informed consent not obtainable
* intubated for more than 3 days
* death within 3 weeks likely
* severe chronic pulmonary disease
* severe chronic cardiac disease
* emergency situation
* intracranial pressure difficult to control
* need for a permanent tracheostoma
* contraindications for dilatative tracheostomy
* severe coagulopathy
* severe respiration difficulties
* intubation/extubation/tube exchange difficulties

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2009-09; Primary Completion 2011-11 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Intensive Care Unit Length of Stay (ICU-LOS) | open
  The primary endpoint is assessed as days from admission to until discharge from the intensive care unit.

SECONDARY OUTCOMES:
Time of ICU-dependence | open
  This secondary endpoint is assessed as days from admission to a pre-defined status that would allow discharge from ICU (absence of active infection, vasopressors, pulmonary and cardial instability etc.)
Functional Outcome | admission, discharge, at 6 months
  This secondary endpoint is assessed as the modified Rankin Scale (mRS) at the above named timepoints.
Mortality | during stay, after 6 months
  This secondary endpoint is assessed as time and type of death during the ICU-stay and 6 months after admission.
Hospital Length of Stay | open
  This secondary endpoint is assessed as days spent at the recruiting hospital from admission to discharge.
Duration of Ventilation | open
  This secondary endpoint is assessed as half-days on the ventilator until the patient is ventilator-independent for 24 h.
Duration and Quality of Weaning | Within ventilation time
  This secondary endpoint is assessed as half-days spent under the possible application of a weaning protocol, and spent within specific phases of such a protocol.
Time of Analgosedation Dependence | within ICU-LOS
  This secondary endpoint is assessed as half-days requiring the application of sedatives and analgesics which are also specified.
Vasopressor Dependence | within ICU-LOS
  This secondary endpoint is assessed as half-days spent under vasopressors.
Time of Antibiotic Treatment | within ICU-LOS
  This secondary endpoint is assessed as half-days under antibiotic treatment
Pneumonias | within ICU-LOS
  This secondary endpoint is assessed as episodes (pre-defined by diagnostic criteria) of pneumonia.
Occurrence and Duration of Sepsis | within ICU-LOS
  This secondary endpoint is assessed as the number of episodes and duration of sepsis as pre-defined by diagnostic criteria.
Number and type of complications associated with the procedure | 10 days post tracheostomy
  This secondary endpoint is assessed as the number and types of complications arelated to tracheostomy (i.e. bleeding, mispositioning, malfunction, replacement demand,etc.).
Cost of Treatment | within ICU-LOS
  This secondary endpoint is assessed as the total ICU-costs etsimated by length of stay and severety-derived DRG-multiplicator of each individual patient.

CONTACTS AND LOCATIONS:
Overall Officials: Bösel Julian, Dr, MD, Principal Investigator — Department of Neurology, University of Heidelberg; Thorsten Steiner, Prof, MD, Study Chair — Department of Neurology, University of Heidelberg
Locations (1):
- NeuroIntensive Care Unit, Department of Neurology, University Hospital Heidelberg, Heidelberg, Germany

REFERENCES:
- [Background] Bosel J, Schiller P, Hook Y, Andes M, Neumann JO, Poli S, Amiri H, Schonenberger S, Peng Z, Unterberg A, Hacke W, Steiner T. Stroke-related Early Tracheostomy versus Prolonged Orotracheal Intubation in Neurocritical Care Trial (SETPOINT): a randomized pilot trial. Stroke. 2013 Jan;44(1):21-8. doi: 10.1161/STROKEAHA.112.669895. Epub 2012 Nov 29. PMID 23204058